CLINICAL TRIAL: NCT05599035
Title: Sleep Disorder in Parkinson Disease and rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: sleep disorder in parkinson
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-01

CONDITIONS: Sleep Disorder; Parkinson Disease
Keywords: sleep disorder Parkinson disease; rTMS
MeSH Terms: conditions — Sleep Wake Disorders; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This study included 30 PD patients and 20 normal volunteers' age and sex matched that were recruited .The diagnosis of PD was done according to UK Brain bank Criteria for diagnosis of PD. Out of them we selected only patients with sleep disturbance according to Self-reported questionnaire for non-motor symptoms (sleep disturbance section; Question 23, 24, 25, 26 as follow 23-Difficulty getting to sleep at night or staying asleep at night 24. Intense, vivid dreams or frightening dreams. 25. Talking or moving about in your sleep as if you are 'acting out' a dream 26. Unpleasant sensations in your legs at night or while resting, and a feeling that you need to move.,) (NMSQuest) or frightening dreams All patients fulfilled by Parkinson's disease sleep scale (PDSS). Treatment was maintained constant during the trial. Each patient under levodopa (Sinemet 250/25; ½ table 3 times per day) and anticholinergic (cogenitol ½ table 3 times per day).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Out of 45 PD patients, 30 patients had sleep disturbance and 6 out of them refused to be participated in the study . Group allocations (active or vs sham with ratio 2 (16 cases):1(8 cases) were placed in serially numbered closed envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1st group received active rTMS, (Active Comparator): Active rTMS was applied using a figure-of-8 coil (7-cm diameter loop) positioned over the parietal area for ten sessions (10 trains, with frequency of stimulation 20-Hz, each lasting for 10 seconds with an inter-train interval of 30 seconds. The intensity of stimulation was set at 80% of the RMT for the first dorsal interosseous (FDI) of the contralateral hand with a total 2000 pulses for each hemisphere). Each patient received five sessions /week for two consecutive weeks with ten total sessions over the parietal area. The parietal region was determined according to the 10-20 system for electroencephalographic electrode positioning at P3 and P4, respectively.
  Interventions: Device: repititive transcranial magnetic stimulation
- 2nd group was the sham group (Sham Comparator): rTMS was applied using the same parameters, but with the coil edge was applied perpendicular to the scalp in the sagittal plane jut to reproduce the noise of the stimulation
  Interventions: Device: repititive transcranial magnetic stimulation

INTERVENTIONS:
Device: repititive transcranial magnetic stimulation — a figure-of-8 coil (7-cm diameter loop) positioned over the parietal area for ten sessions (10 trains, with frequency of stimulation 20-Hz, each lasting for 10 seconds with an inter-train interval of 30 seconds. The intensity of stimulation was set at 80% of the RMT for the first dorsal interosseous (FDI) of the contralateral hand with a total 2000 pulses for each parietal area.)

SUMMARY:
The crude prevalence rate of Parkinson's disease in Upper Egypt governorates ranging from 557-436/100,000 (Assiut and Qena governorates respectively) which was one of the highest prevalence of PD around the world .Parkinson's disease patients report having complaints of disrupted sleep anywhere from 60 to 98 %. This is one of the most common non-motor symptoms, and it is a substantial contributor to the diminished quality of life associated with Parkinson's disease. PD patients have poor sleep maintenance and fragmentation (Comella 2007, Khedr et al. 2013). Khedr et al (2013) found that; 78.6% out of 112 patients with PD had sleep disturbances with the commonest complaint being difficulty getting to sleep at night or staying asleep (46.4%) followed by vivid nightmares and night terrors (27.7%). In other studies, 80-90% of PD patients have had sleep difficulty with virtually all patients having symptoms at some time in the course of the disease .

DETAILED DESCRIPTION:
The pathophysiology of PD sleep problems is unclear. Degeneration of major sleep control centers in the brainstem is a leading factor . In addition to dopaminergic medication, nocturnal akinesia, depression and restless legs syndrome, may contribute to sleep disturbances in Parkinson's disease .Previous studies linked dopaminergic impairment in the hypothalamus to sleep disturbances in PD.

Repetitive transcranial magnetic stimulation (rTMS), non-invasive magnetic stimulation of the cerebral cortex is utilized as non-pharmacological therapy in PD with varying degree of results on the motor symptoms. rTMS has also an impact sleep organization in healthy people both during and before sleep.

The effects of rTMS on sleep have been studied in PD in two previous studies, both of which applied HF over either the motor or parietal cortex. They reported improvement in sleep by subjective and objective measures. However, one of the studies found that the improvement seen on polysomnographic (PSG), the other study found improvement in actigraphic recordings. One sham-controlled trial of the effect of rTMS on sleep in patients with PD also revealed substantial placebo-related improvement on subjective questionnaires (i.e., Parkinson Disease Sleep Scale, Hamilton Depression Rating Scale, Unified Parkinson Disease Rating Scale), with sleep improvement found equally between active and sham stimulation groups . Interestingly, in this trial rTMS showed no changes recorded in actigraphy parameters.

Huang et al. 2018 examined the effect of LF rTMS over the parietal cortex in patients who had generalized anxiety disorder with comorbid insomnia and assessed Hamilton Rating Scale for Anxiety (HRS-A), and PSQI. In their trial, PSQI improvements were seen in active rTMS but not in sham stimulation, making this the second trial of a sham-controlled trial without pronounced placebo effect. Additionally, a positive correlation was seen between improvement in the HRSA anxiety scores and PSQI scores which could suggest that sleep improvement was associated with anxiety improvement. It was not known whether the improvement seen in insomnia and anxiety was independent, and whether rTMS really had an intrinsic role in sleep (Rosenquist and McCall 2019) In another study, Jiang et al. 2013 evaluated the effect of rTMS versus medication versus cognitive behavioral therapy in chronic insomnia. They performed the assessments with PSG and PSQI. Based on PSG findings, rTMS only showed superior improvement in stage 3 and rapid-eye movement sleep.

According to the above mentioned studies rTMS seems to have the ability to improve sleep disorders.

The literature in this area remains scarce, with few randomized clinical trials on rTMS and insomnia. Available studies have found mixed results, with some studies reporting subjective sleep improvement while objective improvement is less consistent.

Despite the significant prevalence of sleep disturbances in PD patients, rTMS's influence on sleep has not been objectively evaluated. To date, the exact mechanism by which rTMS is thought to influence sleep has yet to be fully explained particulary in PD.

The present study aimed to analyse the sleep disturbance in PD patients compared with normal volunteers and to objectively evaluate if rTMS has impact on sleep disorders or not in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PD was done according to UK Brain bank Criteria for diagnosis of PD. Out of them we selected only patients with sleep disturbance All patients fulfilled by Parkinson's disease sleep scale (PDSS).

Exclusion Criteria:

* Patients with PD with disturbed conscious level, severe cognitive impairment, psychosis, and medical problems such as (Renal failure, Liver cell Failure, Respiratory Failure, and endocrinal impairment), patients with other types of Parkinsonism as (Multisystem atrophy, supranuclear palsy, and encephalitic Parkinsonism) and patients had contraindication of magnetic stimulation (metallic piece, pacemaker, epilepsy) were also excluded from the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Parkinson's disease sleep scale (PDSS) | 1 month
  The PDSS is a visual analogue scale addressing 15 commonly reported symptoms associated with sleep disturbance overall quality of night's sleep (item 1); • sleep onset and maintenance insomnia (items 2 and 3); • nocturnal restlessness (items 4 and 5); • nocturnal psychosis (items 6 and 7) • nocturia (items 8 and 9); • nocturnal motor symptoms (items 10-13); • sleep refreshment (item 14); • daytime dozing (item 15).
polysomenography | 1 month
  This polysomnography systematically monitored the electroencephalogram (EEG) (C3-A2, C4-A1), electrooculogram (EOG), electromyogram of the chin (EMG), electrocardiogram (EKG), body positions, nasal and oral airflow, thoracic and abdominal effort, limb movements, pulse oximetry, and snoring sound level.

SECONDARY OUTCOMES:
Beck Depression Inventory | 1 month
  It is a 21-question multiple-choice self-report inventory, one of the most widely used for measurment severity of depression the BDI-II also contains about 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used differ from the original:
  0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression
Unified Parkinson's Disease Rating Scale (UPDRS) | 1 month
  it is a rating scale for assessment of motor and non-motor functions in PD. This assessment included in 4 parts: Part I contains mental section consisting of 4 items (intellectual impairment, thought disorder, depression and motivation), part II consists of activities of daily life with the 12 questions covering many activities like hygiene, dressing, writing and freezing during walking, part III consists of the motor clinical assessment with 14 items (speech, facial expression, tremors at rest, action tremor, rigidity, finger taps, hand movement, rapid alternating movements of hands, leg agility, arising from chair, posture, gait, postural stability, bradykinesia), while part IV is addition of drug complications (dyskinesia, clinical fluctuations). We used motor clinical assessment part III in which each item ranked from 0 (normal), 1 (mildly impaired), 2 (moderately impaired), 3 (severely impaired), 4 (can barely perform the task).
Cognitive assessment using Montreal Cognitive assessment | 1 month
  score 0-30

CONTACTS AND LOCATIONS:
Locations (1):
- Eman Khedr, Asyut, Egypt

REFERENCES:
- [Background] Oerlemans WG, de Weerd AW. The prevalence of sleep disorders in patients with Parkinson's disease. A self-reported, community-based survey. Sleep Med. 2002 Mar;3(2):147-9. doi: 10.1016/s1389-9457(01)00127-7. PMID 14592234
- [Background] Chaudhuri KR, Yates L, Martinez-Martin P. The non-motor symptom complex of Parkinson's disease: a comprehensive assessment is essential. Curr Neurol Neurosci Rep. 2005 Jul;5(4):275-83. doi: 10.1007/s11910-005-0072-6. PMID 15987611
- [Background] Arias P, Vivas J, Grieve KL, Cudeiro J. Double-blind, randomized, placebo controlled trial on the effect of 10 days low-frequency rTMS over the vertex on sleep in Parkinson's disease. Sleep Med. 2010 Sep;11(8):759-65. doi: 10.1016/j.sleep.2010.05.003. Epub 2010 Jul 31. PMID 20674489
- [Background] Khedr EM, Farweez HM, Islam H. Therapeutic effect of repetitive transcranial magnetic stimulation on motor function in Parkinson's disease patients. Eur J Neurol. 2003 Sep;10(5):567-72. doi: 10.1046/j.1468-1331.2003.00649.x. PMID 12940840
- [Background] Khedr EM, Fawi G, Abbas MA, Mohammed TA, El-Fetoh NA, Attar GA, Zaki AF. Prevalence of Parkinsonism and Parkinson's disease in Qena governorate/Egypt: a cross-sectional community-based survey. Neurol Res. 2015 Jul;37(7):607-18. doi: 10.1179/1743132815Y.0000000020. Epub 2015 Mar 23. PMID 25796953
- [Background] Khedr EM, Al Attar GS, Kandil MR, Kamel NF, Abo Elfetoh N, Ahmed MA. Epidemiological study and clinical profile of Parkinson's disease in the Assiut Governorate, Egypt: a community-based study. Neuroepidemiology. 2012;38(3):154-63. doi: 10.1159/000335701. Epub 2012 Mar 29. PMID 22473384
- [Background] Khedr EM, El Fetoh NA, Khalifa H, Ahmed MA, El Beh KM. Prevalence of non motor features in a cohort of Parkinson's disease patients. Clin Neurol Neurosurg. 2013 Jun;115(6):673-7. doi: 10.1016/j.clineuro.2012.07.032. Epub 2012 Aug 16. PMID 22902078